CLINICAL TRIAL: NCT04716296
Title: Intraoperative Use of Ketamine for Awake Deep Brain Stimulation (DBS) Surgery Compared to Standard Procedure
Brief Title: Ketamine in Deep Brain Stimulation (DBS) Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Idit tamit, Head of DBS surgery unit, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0328-20-RMC
Record Dates: First submitted 2020-10-09; First posted 2021-01-20 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2023-03

CONDITIONS: Deep Brain Stimulation
MeSH Terms: interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: blinded: The participant , the neurologist, the neurophysiologist and neuropsychologist treating the participant will be blinded to the randomization arm. The neurosurgeon and anesthesiologist assigned to the patient will be unblinded to the randomization arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine arm (Experimental): Treatment arm consisting of patients randomized to receive a low dose of ketamine for the second stage of DBS surgery.
  Interventions: Drug: Ketamine
- Control arm (Active Comparator): Control arm consisting of patients randomized to receive sham control of saline during the second stage of DBS surgery.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ketamine — Ketamine will be given for the second stage of the DBS surgery.
  Arms: Ketamine arm
Drug: Saline — Saline will be given for the second stage of the DBS surgery.
  Arms: Control arm

SUMMARY:
Deep brain stimulation (DBS) is a well-established and effective treatment for motor symptoms resulting from idiopathic Parkinson's disease (PD). During the DBS surgery , a brain electrode is implanted in the basal ganglia, which is involved in the pathophysiology of the disease. The surgery consists of three steps: 1. Opening the skin, drilling the skull bone and inserting a temporary electrode. 2. Recording electrical activity of the brain, electrical stimulation of the brain which guide the implantation of the electrode.3 Transferring wires and implanting a subcutaneous pacemaker battery in the chest area.

Today, standard treatment protocols consist undergoing the second stage (or first and second stage, depending on the treatment center protocol) of the surgery awake (under local anesthesia only). As systemic anesthetics affect cerebral electrical activity and prevent patient cooperation, they inhibit precise identification of the cerebral target under 'physiological navigation' guided by electrical recording and brain stimulation. As a result, the accuracy of electrode implantation decreases. However, undergoing surgery in an awake format often causes severe patient discomfort and anxiety necessitating shortening the length of surgery or aborting the surgery.

As such there is a need for establishing an alternative anesthesia protocol for DBS surgeries.

Ketamine is considered a unique anesthetic due to its hypnotic properties, analgesia, and possible amnesia. Standard doses of ketamine are currently used worldwide to treat patients with various injuries and brain diseases. Research from monkeys has shown that ketamine (in low dose) does not affect electrical brain activity used for physiological navigation.

The investigators therefore propose a prospective , randomized , blinded study to evaluate the utility of low dose of ketamine in the second stage of DBS surgeries for increasing patient satisfaction and cooperation without detracting from the accuracy of physiological navigation to the cerebral target.

This study will compare two treatment arms :

Treatment arm consisting of patients randomized to receive a low dose of ketamine for the second stage of DBS surgery.

Control arm consisting of patients randomized to receive sham control of saline during the second stage of DBS surgery.

DETAILED DESCRIPTION:
1. On the day before surgery the participant will be shown 10 objects that he should remember. On the day after surgery he will be requested to recall the objects he remembers and to answer the level of anxiety he is feeling using the Visual Anxiety Scale.
2. In the event of discharges (a possible side effect of ketamine due to muscarinic / parasympathetic stimulation), a single dose of scopolamine (1 mg - ) will be given intravenously.
3. At the end of the surgical phase of opening (of the same side being operated on) the propopol will be discontinued (as routinely done), and a continuous low-dose ketamine infusion (0.25 mg per kilogram per hour) will be given until the permanent electrode is implanted on the same operated side, or in the event that unwanted side effects that can't be controlled appear.
4. During surgery, monitoring of muscle activity (EMG) and brain activity (EEG) will be performed
5. During the operation a short canola will be inserted through the meningeal opening and fixed to the surface of the cerebral cortex.

   Through the cannula A 10 mm deep microelectrode will be inserted, which will record electrical activity from the cerebral cortex for several minutes (up to 15 minutes). During the recording period the patient may be asked to perform a simple cognitive task using a computer or iPad. Following the recording the canola and the microelectrode will be removed and the canola will be inserted to the depth of the brain as part of the standard surgery and through it the microelectrode will be inserted into the brain target, and recording of electrical activity from the depths of the brain, as is customary will be performed. At the end of the ketamine phase, at the end of the electrophysiological monitoring required for navigation, prior to the electrical stimulation, when the electrode is placed at the bottom of the sub-thalamic nucleus, the patient will be shown for 60 seconds 10 images of objects (a single object in each image, different from the objects presented to him the day before) which he will asked to remember. At the same time on the screen will present electrical recordings from the depth of the brain (MER) by the brain electrode. In addition, the patient will be asked grade the anxiety level he is experiencing using the Visual Anxiety Scale (VAS) .
6. On the day after surgery, the patient will be asked to recall which objects were presented to him the day before the operation and during the operation. Note that the two object lists will be from a database of objects used in functional day-to-day life (standard lists used for the CMT test - contextual memory test). In addition, the patient will be asked to answer a Visual Anxiety Scale (VAS) and the Iowa satisfaction score questionnaire detailing the patients overall overall experience, mood and feelings during surgery.

   These assessments will be performed by a neuropsychologist and using a validated questionnaire.
7. Two weeks surgery, the patient will be presented with pictures of various objects and will be asked to recall which of them were presented before and during surgery. In addition the patient will be requested to fill grade his VAS anxiety scale and the IOWA questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and above
* Patients with history of Parkinson's disease
* Patients undergoing deep brain stimulation surgery on subthalamic nucleus from the neurology and the neurosurgery at Beilinson hospital
* Patients with the ability to comply with the study requirements and undergoing Patients whom fulfill all above requirements will be approached for enrollment.

Exclusion Criteria:

* Patients who can't cooperate and fulfill study requirements.
* Patients who are at increased risk for performing study related tasks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Electrophysiological recordings MER, Local field potentials and multiunit activity | During surgery
  Efficacy of Ketamine for use of the second stage of DBS surgery

SECONDARY OUTCOMES:
Side effects from ketamine use | During surgery
  Example : hypertension resulting following ketamine use.
The participants neurological status | During surgery
  Participants' neurological status
Patients satisfaction levels measured using owa Satisfaction with Anesthesia Scale | Up to two weeks postoperatively
  Overall participant satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Idit O Tamir, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel